CLINICAL TRIAL: NCT07179224
Title: EEG Monitoring of rTMS-Induced Prefrontal Cortex Reactivity in Various rTMS Stimulation Locations
Brief Title: EEG Changes After rTMS Stimulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTL-699_CTCZ300
Record Dates: First submitted 2025-09-11; First posted 2025-09-17 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Brain Electrical Reactivity to BTL-699-2 Stimulation
Keywords: ExoTMS; EXOMIND; EEG
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment with EXOMIND (BTL-699-2) (Experimental): Transcranial magnetic stimulation with the EXOMIND (BTL-699-2) device
  Interventions: Device: Treatment with EXOMIND (BTL-699-2)

INTERVENTIONS:
Device: Treatment with EXOMIND (BTL-699-2) — Transcranial magnetic stimulation with the EXOMIND (BTL-699-2) device will be delivered across various stimulation locations. The intensity will be carefully adjusted based on subject feedback, but it should not exceed 70% of the motor threshold.
  Other Names: EXOMIND (BTL-699-2) with ExoTMS

SUMMARY:
The goal of this clinical trial is to explore the brain's electrical reactivity, monitored using EEG, following the EXOMIND (BTL-699-2) stimulation across various stimulation locations. The main question it aims to answer is:

What is the brain's cortical electrical reactivity, monitored using EEG, following the EXOMIND (BTL-699-2) stimulation across various stimulation locations?

Participants will be asked to:

* Undergo 1 treatment visit
* Undergo electroencephalography (EEG) measurements
* Complete Therapy Comfort Questionnaires

DETAILED DESCRIPTION:
This is a non-randomized, prospective, single-center, single-arm, open-label, interventional study. All participants will be treated with the EXOMIND (BTL-699-2) device.

Before the first stimulation, a resting EEG recording will be performed for 3 minutes with the subjects' eyes closed and 3 minutes with the subjects' eyes open.

The treatment administration phase consists of one (1) treatment visit. The intensity will be carefully adjusted based on subject feedback, but it should not exceed 70% of the motor threshold.

EEG measurements will be conducted, and the Therapy Comfort Questionnaire will be administered during the treatment visit.

The treatment area will be examined for possible adverse events after the stimulation and during both follow-up visits.

The safety follow-up visits will be 2 weeks (± 2 days) and 1 month (± 5 days) after the treatment visit.

After completing the final follow-up visit (1 month after the treatment visit), the patient's participation in the study will be considered complete. The estimated duration of participation, from the initial visit to the final follow-up, is approximately 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Age > 19 years
* Ability to determine the motor threshold of the participant.
* Willingness to maintain on pre-study psychotherapeutic regime, and prescribed medications at a stable therapeutic dosage for at least 2 months prior to study entry.
* Willingness to comply with study instructions and to return to the clinic for the required visits
* Willingness to undergo EEG examination and proceed with the instructions from the study staff during the measurement
* Women of child-bearing potential are required to use birth control measures during the whole duration of the study

Exclusion Criteria:

* electronic implants (Implanted stimulator devices in or near the head - rTMS devices are contraindicated for use in patients who have active or inactive implants including device leads, deep brain stimulators, cochlear implants, ocular implants, and vagus nerve stimulators, implanted devices such as cardiac pacemakers, defibrillators, and neurostimulators.),
* metallic, ferromagnetic or other magnetic-sensitive implants/objects in or near the head*,
* application in the heart area,
* persons with a tendency to seizure (hypotonic, epileptic),
* ongoing anticoagulation therapy,
* ongoing severe or life-threatening condition,
* ongoing renal dialysis therapy or decompensated** renal insufficiency,
* decompensated* hemorrhagic conditions, blood coagulation disorders, cardiovascular diseases,
* malignant or benign tumour (within 30 cm of the treatment coil),
* fever,
* application over or in the near proximity (within 30 cm of the treatment coil) of tattoos with metallic ink
* pregnancy or nursing
* suicidal tendencies or recent attempt to commit suicide,
* concurrent use of electroconvulsive therapy or vagus nerve stimulation,
* ongoing or recent changes (less than 60 days) in intake doses of any pharmaceutical - products, standalone or in combination, that might lower the threshold of seizure potential,
* ongoing withdrawal conditions from any dependence substance or medication associated with altered seizure risk history,
* a psychotic disorder, including schizoaffective disorder, bipolar disease, or major depression with psychotic features,
* history of primary or secondary tumors in CNS, cerebral aneurysm,
* history of increased intracranial pressure or head trauma with loss of consciousness.
* any medication that may alter EEG report (such as benzodiazepines, barbiturates, carbamazepine, valproate, phenothiazines, clozapine, tricyclic antidepressants, lithium, etc.), any other disease or condition at the investigator discretion that may pose risk to the patient or compromise the study

  * rTMS devices are contraindicated for use in patients who have conductive, ferromagnetic or other magnetic-sensitive metals implanted in their head (with some exceptions in the mouth - standard amalgam dental fillings, single post dental implants, and dental bridge work. When these objects are present monitor the patient during therapy and have the patient notify the operator of warming or other sensation; cease rTMS treatment in event of warming sensation) or within 30 cm of the treatment coil. (Examples include implanted electrodes/stimulators, aneurysm clips or coils, stents, bullet fragments, jewellery, and hair barrettes) **This term applies to patients with a documented medical history of a decompensated health condition requiring medical treatment and/or medication, yet has not received such treatment and/or medication. Patients who use certain medications only for preventive purposes, without any proven previous health condition failure are not considered contraindicated.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-09-17 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of Eletrical Reactivity using EEG | 12 months
  The primary outcome is the comparison of changes in EEG power spectral density (PSD) within specific regions for each stimulation location, as well as a comparison of these results between different stimulation locations. These analyses will be performed across all measured participants. EEG measurement will be performed after the stimulation of each location.

SECONDARY OUTCOMES:
Assessment of Therapy Comfort | 12 months
  Therapy Comfort Questionnaire will be used for evaluating the comfort during the treatment sessions. The Therapy Comfort questionnaire will be administered after the stimulation of each location. Therapy Comfort questionnaire consists of the question "I found the treatment comfortable", to which responses are based on a 5-point Likert scale (1 = "strongly disagree", and 5 = "strongly agree"). A higher score for the statement "I found the treatment comfortable" indicate higher therapy comfort.
Assessment of Pain During Therapy | 12 months
  The Therapy Comfort Questionnaire will be used to evaluate pain experienced during the treatment session. It will be administered after the stimulation of each location. The questionnaire includes a 10-point Numeric Analog Scale for pain (0 = no pain, 10 = worst possible pain). Lower scores on the Numeric Analog Scale indicate lower levels of pain.
Incidence of Treatment-related Adverse Events | 12 months
  Monitoring of adverse reactions and side effects will be performed to identify side effects and adverse events associated with the treatment using the BTL-699-2 device.

CONTACTS AND LOCATIONS:
Locations (1):
- DP Neuro s.r.o., Prague, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No